CLINICAL TRIAL: NCT04488887
Title: Evaluation of the Repeatability and Reproducibility of Different Quantitative Optical Coherence Tomography Angiography Metrics in Retinal Disorders
Brief Title: OCTA Metrics Repeatability and Reproducibility in Different Disorders
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Osama Abdelfattah Sorour, Retina Consultant & the principal investigator, Tanta University
Other Study IDs: 33875/6/20
Record Dates: First submitted 2020-07-24; First posted 2020-07-28 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Diabetic Retinopathy; Myopia; Choroidal Neovascularization; Healthy
MeSH Terms: conditions — Diabetic Retinopathy; Myopia; Choroidal Neovascularization

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Diabetic retinopathy Group: Patients with non-proliferative and proliferative diabetic retinopathy with clear media will be recruited.
  Interventions: Diagnostic Test: Optical coherence tomography angiography
- Myopia Group: Patients with different grades of myopia, with accurate segmentation will be recruited
  Interventions: Diagnostic Test: Optical coherence tomography angiography
- Choroidal neovascularization group: Patients with active choroidal vascularization without scarring will be recruited
  Interventions: Diagnostic Test: Optical coherence tomography angiography
- Healthy controls: Healthy individuals without retinal disorders will be included for comaprison
  Interventions: Diagnostic Test: Optical coherence tomography angiography

INTERVENTIONS:
Diagnostic Test: Optical coherence tomography angiography — patients in all groups will be examined with optical coherence tomography angiography, for every eye 3 macular and 3 papillary scans will be performed by two different OCTA machines, analysis will be carried out to evaluate the repeatability and reproducibility of the test

SUMMARY:
Retinal imaging is a corner stone in diagnosis of most retinal disorders. Standard imaging techniques e.g. fluorescein angiography and color fundus photography have a lot of limitations including limited resolution, invasive nature in cases of fluorescein angiography, and inability to segment the retina, accordingly, and only 2D image is provided.

Optical coherence tomography angiography (OCTA) is a recent noninvasive imaging technique that allows for volumetric visualization of eye vasculature. OCTA has shown promise in better elucidating the pathophysiology of several retinal vascular diseases. Swept-source OCTA uses long wavelength ̰ 1,050nm, which can penetrate through deeper layers of the eye and can traverse opacities of media such as cataracts, hemorrhages and vitreous opacities.

Optical coherence tomographic angiograms can further be manually or automatically segmented with preprogrammed software to highlight individual layers of the retina, optic nerve head choriocapillaris, and choroid. The user can either analyze en face images extending from the inner limiting membrane to choroid or use automated views to locate a vascular or structural lesion within the retina.

Different quantitative metrics has been extracted from enface OCTA images including vessel density, FAZ area, choriocapillaries flow deficit, intercapillary area and fractal dimension. These metrics are helpful in evaluation the retinal perfusion and used by physicians to assess various retinal vascular disorders.

Although some previous literatures had discussed the repeatability of OCTA metrics, however, comprehensive evaluation of widely used metrics in various retinal condition has not be done. Additionally, recent data suggest that various methods of calculation of these metrics my yield final different results of the same metric.

DETAILED DESCRIPTION:
This will be prospective cross-sectional study. This research will be done in the period between 1 August and 31 December 2020 and will include 80 eyes from patients with following disorders:

Group 1: Patients with diabetic retinopathy Group 2: Patients with myopia Group 3: patients with choroidal neovascularization Group 4: control eyes with no retinal disease. Inclusion criteria: Patients above 18 years in age with any of above retinal condition and clear media allowing for imaging will be included.

Exclusion criteria will include; Maculopathies (hereditary or acquired), optic nerve head pathologies (tilted disc, drusen, optic disc edema, atrophy, etc.), optic neuropathies (demyelinating, infectious, ischemic, etc.), adjusted IOP for central corneal thickness more than 21 mmHg, surgery-induced corneal edema and dense cataracts that can disrupt images, history of vasoactive agents (calcium antagonists, nitric oxide, etc.) use, systemic diseases (vasculitis, diabetes mellitus, hypertension, etc.) and any previous ocular surgery, patients with bad quality images or complicated surgeries will be excluded.

All patients will be subject to Full ophthalmologic examination and OCTA imaging. High-quality 3 x 3 mm and 6 x 6 mm OCTA macular scans and 4.5 × 4.5-mm papillary scan with strong signal-noise ratio and adequate centration on the fovea and optic nerve head respectively will be selected.

For each patient 10 successive scans will be generated to allow for the analysis of repeatability. Patient will be imaged in the same day at two different OCTA devices Dri Triton (Topcon, Japan) and Cirrus OCT (Zeiss, USA) to investigate the reproducibility of the measurements.

Automated segmentation will be used to evaluate superﬁcial and deep capillary retinal plexus projections. If errors in segmentation were detected, manual correction would be performed. The superﬁcial retinal capillary plexus (SCP) was delineated with an inner boundary at the internal limiting membrane (ILM) and an outer boundary 10 µm inside the inner plexiform layer (IPL). The deep retinal capillary plexus (DCP) was segmented with an inner boundary 10 µm inside the IPL and an outer boundary at 10 µm beneath the outer plexiform layer (OPL). In addition, the total retinal capillary plexus (TCP) was manually customized by selecting the inner boundary at the ILM and the outer boundary set at 40 µm above the retinal pigment epithelium (RPE) to avoid any ﬂow signals from choriocapillaries.

We will evaluate the following metric from enface OCT angiogram; vessel density, vessel density, intercapillary area, fractal dimension and skeletonized vessel density.

Every included patient in this study will have unique code number referring to the file where all his data will be kept confidential. Only macula and optic disc will be imaged. Additionally, patients' personal data will be hidden during using of these images. All patients' data will be used for scientific research only and will be kept totally confidential. Comprehensive explanation of all aspects of this study will be given to patients before their participation in it, an informed consent will be obtained from the patients before their enrolment in the study. Although no documented adverse effects from OCTA imaging on the patients to date, however, any unexpected risks appeared during the research will be cleared to the participants and the ethical committee on time.

Statistical analysis will be performed using SPSS software (version 25; SPSS, Inc., Chicago, IL, USA). the intraclass correlation coefficient (ICC) and coefficient of variation (CV) will be calculated. ICC is the correlation between two variables measured at the same time point, with values ranging from 0 to 1 (<0.40, poor; 0.40-0.59, fair; 0.60-0.74, good; 0.75-1.00, excellent). The CV (%) will be calculated as 100 × standard deviation/overall mean, and a value <10% represents good repeatability of the measurement.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or above, that fall in any of the study groups
* Clear media allowing for imaging

Exclusion Criteria:

* Maculopathies (hereditary or acquired)
* Optic nerve head pathologies (tilted disc, drusen, optic disc edema, atrophy, etc.)
* Optic neuropathies (demyelinating, infectious, ischemic, etc.),
* corneal edema and dense cataracts that can disrupt images
* history of vasoactive agents (calcium antagonists, nitric oxide, etc.)
* systemic diseases (vasculitis, diabetes mellitus, hypertension, etc.)
* Previous ocular surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Repeatability and reproducibility of the different OCTA metrics will be carried out in the following disorders; diabetic retinopathy, myopia, choroidal neovascularization, and in healthy controls for comparison.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
The intraclass correlation coefficient (ICC) | 5 months
  ICC is the correlation between two variables measured at the same time point, with values ranging from 0 to 1 (<0.40, poor; 0.40-0.59, fair; 0.60-0.74, good; 0.75-1.00, excellent).
coefficient of variation (CV) | 5 months
  The CV (%) will be calculated as 100 × standard deviation/overall mean, and a value <10% represents good repeatability of the measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Osama A Sorour, MD, Principal Investigator — Tanta University
Locations (1):
- Ophthalmology Department, Faculty of medicine, Tanta Univeristy, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mehta N, Liu K, Alibhai AY, Gendelman I, Braun PX, Ishibazawa A, Sorour O, Duker JS, Waheed NK. Impact of Binarization Thresholding and Brightness/Contrast Adjustment Methodology on Optical Coherence Tomography Angiography Image Quantification. Am J Ophthalmol. 2019 Sep;205:54-65. doi: 10.1016/j.ajo.2019.03.008. Epub 2019 Mar 15. PMID 30885708
- [Background] Byon I, Alagorie AR, Ji Y, Su L, Sadda SR. Optimizing the Repeatability of Choriocapillaris Flow Deficit Measurement From Optical Coherence Tomography Angiography. Am J Ophthalmol. 2020 Nov;219:21-32. doi: 10.1016/j.ajo.2020.05.027. Epub 2020 May 23. PMID 32454035